CLINICAL TRIAL: NCT01651572
Title: Assessment of Post-operative Residual Curarization (PORC) Incidence in Patients Undergoing Surgery With General Anaesthesia; Comparison Between Cisatracurium and Rocuronium. A Randomised, Single-blind Phase 4 Study.
Brief Title: Comparison Between Cisatracurium and Rocuronium in Terms of Recovery of the Muscular Strength in the Postoperative Phase After Surgery and General Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Dr. Paolo Feltracco, Principal Investigator, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2633Pbis; 2012-002398-68 (EudraCT Number); CURARI_2012 (Other: Comitato Etico dell'Azienda Ospedaliera di Padova)
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Postoperative Residual Curarization; Residual Neuromuscular Block
Keywords: Postoperative residual curarization; Residual neuromuscular block; Complications; Postoperative; Neuromuscular function; Neuromuscular block
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — cisatracurium; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisatracurium (Experimental): Induction and maintaining of anaesthesia with Propofol. Analgesia either with Fentanyl or Fentanyl+Remifentanyl.
  Cisatracurium (Nimbex):
  * initial dose: 0.2 mg/kg
  * maintaining dose: 0.1 mg/kg (repeated anytime TOF-count reaches 2 twitches)
  At the end of the surgical operation, patients will be administered Neostigmine 0.04 mg/kg and Atropine 0.02 mg/kg.
  Patients will be extubated with a TOF-Ratio of at least 0.90.
  Interventions: Drug: Cisatracurium
- Rocuronium (Experimental): Induction and maintaining of anaesthesia with Propofol. Analgesia either with Fentanyl or Fentanyl+Remifentanyl
  Rocuronium (Esmeron):
  * initial dose: 0.6 mg/kg
  * maintaining dose: 0.15 mg/kg (repeated anytime TOF-count reaches 2 twitches)
  At the end of the surgical operation, patients will be administered Neostigmine 0.04 mg/kg and Atropine 0.02 mg/kg.
  Patients will be extubated with a TOF-Ratio of at least 0.90.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Cisatracurium — Cisatracurium (Nimbex):
  * initial dose: 0.2 mg/kg
  * maintaining dose: 0.1 mg/kg (repeated anytime TOF-count reaches 2 twitches)
  Arms: Cisatracurium
Drug: Rocuronium — Rocuronium (Esmeron):
  * initial dose: 0.6 mg/kg
  * maintaining dose: 0.15 mg/kg (repeated anytime TOF-count reaches 2 twitches)
  Arms: Rocuronium

SUMMARY:
The purpose of this study is to determine the incidence of post-operative residual curarization in our patients and to determine if Cisatracurium and Rocuronium behave differently from each other in terms of residual curarization.

ELIGIBILITY:
Inclusion Criteria:

* general anaesthesia with need to use of neuromuscular-blocking agents
* awakening and extubation of the patient in the operating room and permanence in the PACU for at least 60 minutes
* age 18-80
* surgical operations lasting at least 1 hour
* ASA class I-III
* possibility to apply TOF-monitoring with thumb-acceleromyography
* women of childbearing age not using contraceptives
* women of childbearing age using contraceptives

Exclusion Criteria:

* subjects unable to give a valid consent
* patients in emergency situations
* patients not awakened and not extubated in the operating room
* age above 80 years or under 18 years
* surgical operations lasting less than an hour
* ASA class IV
* impossibility to apply and/or perform TOF-monitoring
* neuromuscular diseases
* intake of therapies interfering with the neuromuscular function
* patients having contraindications for either studied drug
* pregnant women
* women who are breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of PORC | Participants will be followed for the duration of their stay in the post-anaesthesia care unit (PACU), an expected average of 60 minutes.
  To determine the incidence of post-operative residual curarization in our operating rooms, comparing two different neuromuscular-blocking agents: Cisatracurium and Rocuronium.
  The primary endpoint is quantified with TOF-Ratio, determined with the device TOF-Watch SX (Organon, Netherlands). A TOF-Ratio<0.90 defines PORC.
  Three clinical parameters (head-tilt for 5 seconds, ability to swallow, presence of diplopia) are also evaluated.
  TOF-Ratios, as long as the above-mentioned clinical parameters are determined and evaluated at 15, 30 and 60 minutes after extubation of the patient.

SECONDARY OUTCOMES:
Incidence of PORC - comparison between Cisatracurium and Rocuronium | Participants will be followed for the duration of their stay in the post-anaesthesia care unit (PACU), an expected average of 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ori, Prof. M.D., Study Chair — Università degli Studi di Padova - Azienda Ospedaliera di Padova; Paolo Feltracco, M.D., Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Padova, Italy